CLINICAL TRIAL: NCT05247112
Title: Prevalence and Trends of Antimicrobial Resistance of Helicobacter Pylori in Korea
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1504-294-305
Record Dates: First submitted 2022-01-18; First posted 2022-02-18 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori Associated Gastrointestinal Disease; Helicobacter Pylori Infection, Susceptibility to; Helicobacter Pylori 23S rRNA Clarithromycin Resistance Mutation
Keywords: eradication; rescue therapy; antibiotics; resistance; Helicobacter pylori

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — H. pylori strains isolated by study subjects.
  Susceptibility is investigated for each of the H. pylori strains, and mutations (e.g., 23SrRNA, gyrA, etc.) that can decisively cause resistance can be investigated only if necessary. All consent to these biosamples will be obtained in advance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess antimicrobial resistance rates and minimal inhibitory concentrations in H. pylori isolated from patients with upper gastrointestinal disease with long-term period.

DETAILED DESCRIPTION:
Failure of eradication treatment against Helicobacter pylori (H. pylori) is mainly caused by antimicrobial resistance. However, there is no relevant studies have been conducted on the prevalence and trend of antimicrobial resistance, which is considered to have a major determinant of eradication failure. In addition, studying the trend of resistance rate is an important basis for establishing an appropriate strategy for eradication treatment in the future.

Patients who had H. pylori colonies isolated from culture were consecutively enrolled from 2003. From each patient, 1 to 10 H. pylori isolates were isolated. Trends in MIC distribution and prevalence of resistance were investigated for each antimicrobial agent according to time period. Antimicrobi resistances suspected to related with failure of empirical PPI triple, quadruple, and rescue fluoroquinolone-containing treatment were also investigated. Multiple resistance, which is simultaneously resistant to various antibiotics, will also be investigated. Risk factors for the antibiotic resistance will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had a H. pylori infection and had consented to undergo culture analysis via endoscopic resection, in order to determine the minimal inhibitory concentration (MIC) of various antibiotics.

Exclusion Criteria:

* Patients with a concurrent critical illness, who abused drugs or alcohol, who were pregnant or nursing, or those who had received antibiotics, PPIs, or bismuth salts within 4 weeks, were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects of this study all had H. pylori infection. None of them should meet the exclusion criteria. Even though successfully proven H. pylori infection, culture procedures must be successful and the susceptibility must be clearly determined by obtaining MIC values to be finally included in this study. According to the literature, culture is successful at approximately 2/3. Informed consent will be obtained from all study subjects.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Resistance rate | through study completion, an average of 1 year
  It means resistance to an antimicrobial agent applicable for H. pylori eradication. Minimal inhibitory concentration test was performed for amoxicillin, clarithromycin, metronidazole, tetracycline, rifabutin, levofloxacin, and moxifloxacin using agar dilution method.
Minimal inhibitory concentration (MIC) distribution | through study completion, an average of 1 year
  The concentration of specific antibiotics that can kill 50% of H. pylori is defined as MIC50. Each analyzes the ratio of strain according to the concentration of antibiotics.
Multiple resistance, prevalance and trends | through study completion, an average of 1 year
  It is defined as the case where the H. pylori strain shows resistance to several antimicrobial agents at the same time. Multiple resistance is calculated by calculating the proportion of strains with simultaneous resistance to 1> clarithromycin and metronidazole, 2> clarithromycin and fluoroquinolone, and 3> clarithromycin, fluoroquinolone, and metronidazole.

SECONDARY OUTCOMES:
Risk factor for eradication failure or success | through study completion, an average of 1 year
  Risk factors for eradication failure or success could be found in the demographic profile of the study subject along with resistance/non-resistance to each antibiotic to H. pylori and its strain.
  According to previous studies, risk factors related with eradication failure or success are usually known from demographic data such as age, sex, and history of eradication treatment. In our study, we use logistic regression analysis to find out whether these factors have significance.

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph.D, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JW, Kim N, Choi SI, Jang JY, Song CH, Nam RH, Lee DH. Prevalence and trends of multiple antimicrobial resistance of Helicobacter pylori in one tertiary hospital for 20 years in Korea. Helicobacter. 2023 Feb;28(1):e12939. doi: 10.1111/hel.12939. Epub 2022 Dec 7. PMID 36478622